CLINICAL TRIAL: NCT03408249
Title: IBDoc® Canadian User Performance Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bühlmann Laboratories AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IBDoc_UserPerfomance006
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's disease, ulcerative colitis, fecal calprotectin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBD patients (Experimental): IBD patients performing IBDoc calprotectin test and ease-of-use questionnaires
  Interventions: Diagnostic Test: IBDoc calprotectin test; Other: questionnaire

INTERVENTIONS:
Diagnostic Test: IBDoc calprotectin test — Patients are asked to perform a single IBDoc calprotectin home test.
Other: questionnaire — Patients evaluate the ease-of-use of the test, clearness of test results and comprehensiveness of the instructions for use through a specific questionnaire implementing Likert scales.

SUMMARY:
The objective of the IBDoc® user performance evaluation is to demonstrate the ease-of-use of the IBDoc® calprotectin home test to allow patients with inflammatory bowel disease (IBD) to independently and correctly determine calprotectin concentration in their own stool sample. The study is based on Chapter 8 of the International Organization for Standardization (ISO) Standard, ISO 15197:2013 "In vitro diagnostic test systems - Requirements for blood-glucose monitoring systems for self-testing in managing diabetes mellitus". The study is a prospective, multicenter study, not blinded for patients, and includes a total of 61 patients.

DETAILED DESCRIPTION:
The patient will determine the calprotectin concentration in their own stool sample using the IBDoc® assay. For this, the patient will collect a stool sample in a standard collection tube at home. The patients will return to the clinical site with the specimen, where they will receive a standardized IBDoc® training. They will also be given opportunity to perform an IBDoc® practice test using the collected sample. The patients will then perform the full IBDoc® assay using the collected stool sample under the observation of the healthcare provider, who will assess their performance. The final result - the interpretation of the IBDoc® lateral flow assay by the CalApp® smartphone application, to yield a final μg/g calprotectin concentration in stool, will be sent to the health care provider (HCP) via the IBDoc® Web Portal.

The usability of the IBDoc® test will be evaluated according to the following factors:

- Trueness/ accuracy - the patients' ability to obtain correct results will be evaluated by comparing patients' IBDoc® results with reference measurements from the same stool sample using the BÜHLMANN fCAL® ELISA, performed at a laboratory site. For reference measurements the HCP at the clinical site will obtain 3 CALEX® Cap extracts from the patient's stool sample, which will be stored frozen and shipped to the laboratory site.

To exclude bias or inaccuracy that may arise from the analytical performance characteristics of the IBDoc® assay itself, a comparative IBDoc® assay will be performed according to the instructions for use, with the patients' samples in a laboratory. For the comparative IBDoc® measurement the HCP at the clinical site will obtain one CALEX® Valve extract from the patient's stool sample, which will be stored frozen and shipped to the laboratory site.

-IBDoc® Calprotectin test usability, clearness of obtained result, and comprehensiveness of the Instruction for Use will be assessed in the following ways:

* Patient's questionnaire
* HCP's questionnaire - human factors evaluation

The ability of patients to correctly collect and extract stool samples using the CALEX® Valve device will be analysed as an additional module within the IBDoc® User Performance Evaluation. The CALEX® Valve extracts obtained by the patients as part of the IBDoc® procedure will be stored frozen and shipped to the laboratory site. Calprotectin levels in the patients' CALEX® Valve extracts will be determined with the BÜHLMANN fCAL® ELISA and compared to calprotectin reference values obtained from the same stool samples by the HCP's.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 12 years
* IBD Outpatients from a tertiary gastroenterological health care center willing to participate.
* Patients diagnosed with Ulcerative Colitis (UC) or Crohn's disease (CD), according to classical criteria (laboratory testing and exclusion of other possible causes: complete blood count, comprehensive metabolic panel, serological markers e.g. antineutrophil cytoplasmic antibody (ANCA), inflammatory markers in blood and serum: erythrocyte sedimentation rate, C-reactive protein (CRP); fecal occult blood and fecal calprotectin assays; confirmation by endoscopy, histology of a biopsy)
* At least 30% patients should display active disease. This can be defined by a Harvey-Bradshaw index (HBI) > 5 in CD and a clinical Mayo score > 2 in UC
* Remaining patients in clinical remission or only mildly active disease defined by a HBI<7 in CD and a clinical Mayo score < 3 in UC with a stable medical treatment
* In case of a prescribed endoscopy, the observation period starts >3 days after colonoscopy
* Stable care of a treating physician
* Signed informed consent

Exclusion Criteria:

* Other known pathology or predisposition that may interfere with the ability to perform the measurement procedures or that may influence calprotectin levels such as acute diarrhea or chronic use of non-steroidal anti-inflammatory drugs
* Inability to understand the procedures
* Inability to psychologically handle potential test outcomes

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Trueness/ accuracy of patients IBDoc® results | 24 hours
  Patients' IBDoc results are compared to reference calprotectin values obtained by laboratory methods
Quantifiable feedback from the enrolled patients about the ease-of-use of the test | 24 hours
  Ease-of-use of the test, clearness of test results and comprehensiveness of the instructions for use is assessed in a questionnaire, with 12 statements, scored on a 1-to-5 Likert scale, with one (1) indicating "I strongly disagree" and five (5) "I strongly agree". The mean and standard deviation of scores obtained from all participating patients will be evaluated for each statement.
Quantifiable feedback from healthcare providers | 24 hours
  Quantifiable feedback from the healthcare providers about the ability of the patients to correctly perform the IBDoc® assay. Assessment will be made through a questionnaire with five (5) statements, scored on a 1-to-5 Likert scale, with one (1) indicating "I strongly disagree" and five (5) "I strongly agree". The mean and standard deviation of scores obtained from all participating healthcare providers will be evaluated for each statement.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Rosenfeld, MD, Principal Investigator — GIRI (GI Research Institute), Vancouver, Canada
Locations (3):
- Canada (3):
  - Division of Gastroenterology, Department of Medicine, Faculty of Medicine University of Alberta,, Edmonton, Alberta
  - GIRI (GI Research Institute), Vancouver, British Columbia
  - Hôtel-Dieu de Lévis,, Lévis, Quebec

REFERENCES:
- [Derived] Moore AC, Huang VW, Bourdages R, Fedorak RN, Reinhard C, Leung Y, Bressler B, Rosenfeld G. IBDoc Canadian User Performance Evaluation. Inflamm Bowel Dis. 2019 May 4;25(6):1107-1114. doi: 10.1093/ibd/izy357. PMID 30535387